

# STATISTICAL ANALYSIS PLAN

# A randomised study of interferon-free treatment for recently acquired hepatitis C in people who inject drugs and people with HIV co-infection

| Study Title: | A randomised study of interferon-free treatment for recently |
|---|---|
| | acquired hepatitis C in people who inject drugs and people with |
| | HIV co-infection |
| Name of Study Drug: | sofosbuvir/velpatasvir |
| Protocol Number: | VHCRP1401 |
| Protocol Version: | 5.0 |
| Protocol Date: | 4 June 2019 |
| Co-ordinating Principal Investigators: | A/Professor Gail Matthews |
| Name/s of Sponsor: | UNSW Sydney |
| Analysis Type: | Primary – SVR12 |
| Analysis Plan Version: | Final V1.0 |
| Analysis Plan Date: | September 2019 |
| Analysis Plan Author: | Kathy Petoumenos |

# Contents

| LIST OF ABBREVIATIONS | 3 |
|--------------------------------------------------------------|----|
| STUDY DEFINITIONS | 4 |
| STUDY DESIGN AND OBJECTIVES | 5 |
| Study Objectives | 5 |
| Hypothesis | 5 |
| Study design (Figure 1) | 5 |
| Sample size and power | 6 |
| TYPE OF ANALYSIS | 7 |
| Data Safety and Monitoring Board (DSMB) Analysis | 7 |
| Primary analysis: Post-treatment week 12 | 7 |
| GENERAL CONSIDERATIONS FOR DATA ANALYSES | 8 |
| Statistical Methods | 8 |
| Analysis Sets | 8 |
| Data Handling Conventions | 9 |
| Missing Data | 9 |
| Outliers | 9 |
| Data Handling Conventions and Transformations | 10 |
| Visit Windows | 10 |
| Definition of Study Day | 10 |
| Analysis Windows | 10 |
| PARTICIPANT DISPOSITION | 12 |
| Recruitment | 12 |
| Participant Enrolment and Disposition | 12 |
| Protocol violations | 12 |
| BASELINE DATA | 16 |
| Demographic Data and Baseline Characteristics (Table 7 - 11) | 16 |
| STUDY ENDPOINTS | 22 |
| Primary efficacy endpoint | 23 |
| Secondary efficacy endpoints | 23 |
| Virological endpoints (Table 13 and 14) | 23 |
| Primary safety endpoints | 23 |
| Adherence | 23 |
| Other secondary outpoints | 26 |
| SAFETY ANALYSES | 28 |
| Extent of Exposure | 28 |
| Adverse Events | 28 |

| Adverse Event Severity | |
|----------------------------------------------|----|
| Relationship of Adverse Events to Study Drug | 28 |
| Summaries of Adverse Events and Deaths | 28 |
| Serious adverse events (SAE) | 29 |
| Laboratory Evaluation | 29 |

#### LIST OF ABBREVIATIONS

AE adverse event

ALT alanine aminotransferase
APRI AST:platelet ratio index

APTT activated partial thromboplastin time

AST aspartate aminotransferase

BLoQ below the lower limit of quantitation

CI confidence interval
CPT Child-Pugh-Turcotte
DAA direct acting antiviral
ECG electrocardiogram

eCRF electronic case report form

EOT end of treatment FDC fixed-dose combination

FU follow-up
GT genotype
HCV hepatitis C virus
HLGT high level group term
HLT high level term

INR international normalized ratio of prothrombin time

LLOQ lower limit of quantitation

LLT lower level term

LSM liver stiffness measurement

MedDRA Medical Dictionary for Regulatory Activities

MELD Model for End-Stage Liver Disease

PT preferred term Q1 first quartile Q3 third quartile

SAE serious adverse event
SAP statistical analysis plan
SD standard deviation
SOC system organ class

SVR sustained virologic response

SVRx sustained virologic response x weeks after stopping study drug

TD target detected
TND target not detected
ULN upper limit of normal

#### STUDY DEFINITIONS

*HCV virological suppression* is defined as HCV RNA below the lower limit of quantitation (LLoQ) (target not detected [TND] or target detected, not quantifiable [TDnq]).

An end-of-treatment response (ETR) is defined as plasma HCV RNA below the LLoQ (TND or TDnq) at the end of treatment.

Sustained virological response at 4 weeks post-treatment (SVR4) is defined as plasma HCV RNA below the LLoQ (TND or TDnq) at 4 weeks post cessation of treatment.

Sustained virological response at 12 weeks post-treatment (SVR12) is defined as plasma HCV RNA below the LLoQ (TND or TDnq) at 12 weeks post cessation of treatment.

Sustained virological response at 24 weeks post-treatment (SVR24) is defined as plasma HCV RNA below the LLoQ (TND or TDnq) at 24 weeks post cessation of treatment.

*HCV virologic failure* is defined as *non-response* (failure of virological suppression on-treatment with quantifiable HCV RNA at all time points between baseline and end of treatment)

*Reinfection* is defined by the presence of quantifiable HCV RNA after an ETR and detection of infection with an HCV strain that was distinct from the primary infecting strain (heterologous virus on sequencing of Core-E2 and/or NS5B regions).

Relapse is defined by recurrent viraemia by SVR12 where reinfection is not confirmed.

The presentation of recent HCV infection at the time of diagnosis is classified as either acute clinical or asymptomatic infection. Acute clinical infection includes participants with a documented clinical history of symptomatic seroconversion illness (including, but not limited to, the presence of jaundice, nausea/vomiting, abdominal pain, fever and hepatomegaly) and those without clinical symptoms but with a documented peak ALT >10 times the upper limit of normal (ULN) within the 12 months prior to diagnosis. Asymptomatic infection includes participants with anti-HCV antibody seroconversion but no acute clinical symptoms or documented peak ALT <10x ULN.

The duration of HCV infection at screening and baseline will be calculated from the estimated date of infection. The estimated date of clinical infection is calculated as six weeks before onset of seroconversion illness or six weeks before the first ALT >10x ULN. The estimated date of asymptomatic infection is calculated as the midpoint between the last negative anti-HCV antibody or HCV RNA and the first positive anti-HCV antibody or HCV RNA. For participants who were anti-HCV antibody negative and HCV-RNA positive at screening, the estimated date of infection is six weeks before enrolment, regardless of symptom status.

On-treatment adherence will be calculated by subtracting the number of missed doses from the total number of doses prescribed for therapy duration and dividing by the total number of doses prescribed for therapy duration. By pill count and self-reported questionnaire, compliance with sofosbuvir/velpatasvir will be individually calculated at the 80, 90 and 100 adherence levels, defined as receipt of  $\geq 80$ ,  $\geq 90$  or 100% of scheduled doses.

#### STUDY DESIGN AND OBJECTIVES

#### **Study Objectives**

#### Primary objective

The primary objective is to evaluate the proportion of patients with HCV RNA below the level of quantitation (target not detected [TND] or target detected, not quantifiable [TDnq]) at 12 weeks post end of treatment (SVR12) following sofosbuvir/velpatasvir therapy for 6 weeks (short treatment duration) as compared with 12 weeks (standard treatment duration) in people with recent HCV infection (duration of infection ≤12 months).

#### Secondary objectives

- To evaluate the proportion of participants with HCV RNA below the level of quantitation (TND or TDnq) at the end of treatment (ETR), 4 weeks after treatment completion (SVR4) and 24 weeks after treatment completion (SVR24);
- To evaluate the proportion of participants with undetectable HCV RNA through 2 years post treatment;
- To evaluate the levels of adherence, factors associated with suboptimal adherence including HIV status, and the impact of suboptimal adherence on therapeutic response;
- To evaluate the impact of treatment on illicit drug use, injecting behaviour and sexual risk taking behaviour (behavioural survey) during treatment;
- To evaluate safety and tolerability;
- To evaluate the change in HIV RNA and CD4 (on-treatment and end of treatment);
- To evaluate the rate and risk factors for reinfection during and up to 2 years following treatment;
- To evaluate the immunological factors associated with treatment induced clearance and reinfection;
- To evaluate patient interest and attitudes towards long acting parenteral hepatitis C therapy (Long-Acting Hepatitis C Therapy Questionnaire).

#### **Hypothesis**

Six weeks treatment with sofosbuvir/velpatasvir is non-inferior to twelve weeks treatment with sofosbuvir/velpastavir as assessed by sustained virological response at 12 weeks post treatment in the intention-to-treat population (SVR12).

#### Study design (Figure 1)

This is an open label multicentre study. The study consists of a screening phase, treatment phase and follow-up phase to evaluate treatment response and reinfection. Participants will be required to wait a minimum of four weeks form screening before commencing treatment to assess for spontaneous clearance. The maximum wait period allowed between screening and baseline is 12 weeks.



Figure 1: Study Schema

#### Sample size and power

The primary objective of this trial is to establish the non-inferiority of short duration treatment (6 weeks) to the standard duration treatment (12 weeks). Assuming an expected SVR of 90% in the control arm, 113 participants per arm will be required to give 80% chance that the two-sided confidence interval of the difference between regimens has a lower limit greater than -12%.

A total of 250 subjects enrolled and randomised will comprise the intention-to-treat (ITT) population and will form the study population for evaluation of the primary and secondary endpoints.

#### **TYPE OF ANALYSIS**

This document describes the primary statistical analysis for REACT study in accordance with protocol version 5.0.

#### **Data Safety and Monitoring Board (DSMB) Analysis**

This study has a DSMB to review the progress and safety of the study. The DSMB conducted an interim safety and adherence analysis when the first 50 participants had either reached post-treatment week 12 or dropped out of the study and then when a further 10 per arm reached 12 weeks post treatment. At the second review the DSMB recommended termination of the short arm of the study due to inferiority. At the stage of the DSMB recommendation, at total of 196 participants had been randomised, 192 had completed their randomised treatment, a further 4 were randomised to receive 6 weeks and extended to 12 weeks. Therefore, the primary analysis population will be based on 192 participants (99 in standard Arm, and 93 in shortened arm).

#### Primary analysis: Post-treatment week 12

The analysis for the primary endpoint, SVR12, will be conducted after all participants have completed the post-treatment week 12 visit or prematurely discontinue from study. All the safety and efficacy data through to the post-treatment week 12 visit will be cleaned, finalised, and included for the analysis.

# **GENERAL CONSIDERATIONS FOR DATA ANALYSES**

#### **Statistical Methods**

Analysis results will be presented using descriptive statistics. For categorical variables, the number (n) and percentage of participants in each category will be presented. For continuous variables, the number of participants (n), mean and standard deviation (SD), median, interquartile range (IQR, Q1-Q3), range (minimum, maximum) will be reported; for inclusion in the manuscript, an appropriate determination will be made depending on the variable, size and distribution of the population studied.

Statistical tests will be 2-sided and performed at the 5% significance level unless specified.

For all efficacy endpoints, means and proportions with two-sided 95% confidence intervals (CI) will be determined. For the analysis of categorical outcomes, Chi-squared tests or exact equivalents (for small numbers) will be used. For comparison of continuous measures, t tests or non-parametric equivalents will be used as appropriate for the observed data distribution. Changes in injecting behaviour between screening, end of treatment and post-treatment week 12 will be compared using the McNemar test (exact binomial probability).

#### **Analysis Sets**

Analysis sets define the subjects to be included in an analysis. The number of participants eligible for each analysis set will be provided. Participants who were excluded from each analysis set will be summarised, with reasons for exclusion.

#### **Full Analysis Set (ITT population)**

The FAS includes all enrolled participants who were randomised. This will be the analysis set used for the primary efficacy and safety endpoints. Following the DSMB recommendation to cease the study, the primary analysis population will be based on 192 participants (99 in standard Arm, and 93 in shortened arm).

#### **Modified Full Analysis Set**

The modified Intention to Treat (mITT) population includes participants in the FAS excluding those with non-virological reasons for treatment failure (i.e., death, loss to follow up) and reinfection. Participants with confirmed reinfection after achieving an ETR, but prior to the primary efficacy endpoint (SVR12), will be excluded from the mITT.

#### **Per-protocol Analysis Set**

The PP population is defined as all participants who received >90% of scheduled treatment for >90% of the scheduled treatment period with follow-up virologic data to SVR12.

#### **Safety Population**

The Safety population includes all participants who randomised and will be analysed and presented according to the actual on-treatment monitoring arm received during the study.

The ITT population will be used for primary efficacy analyses, and the safety population will be used for all safety analyses.

# Data Handling Conventions Missing Data

For the analyses of categorical HCV RNA data, missing post-treatment HCV RNA data will have the missing data imputed. Missing on-treatment HCV RNA will have the missing data imputed up to the time of the last dose.

If a data point is missing and is preceded and followed in time by values that are "<LLOQ, TND," then the missing data point will be set to "<LLOQ, TND."

If a data point is missing, and preceded and followed by values that are "<LLOQ, target detected," or preceded by "<LLOQ, target detected" and followed by "<LLOQ, TND," or preceded by "<LLOQ, TND" and followed by "<LLOQ, target detected," then the missing value will be set to "<LLOQ, target detected."

If a data point is missing, and preceded and followed by values that are ">LLOQ, target detected," or preceded by ">LLOQ, detected" and followed by "<LLOQ, target detected" or "<LLOQ, TND", then the missing value will be set to ">LLOQ, target detected."

The following scenarios describe a framework for analysis of the primary endpoint based on various anticipated events for the ITT and mITT population:

- i. In the event of the participant dying or becoming lost to follow-up prior to SVR
   12, the participant will be considered to have failed treatment (loss to follow up = failure)
- ii. If the SVR 12 time-point measure is missing, then the next available measure (i.e., SVR 24 or later) will be used. If no future time points are available, the participant will be considered a treatment failure.

Where appropriate, safety data for subjects who did not complete the study will be included in summary statistics.

#### For example:

- If a participant took at least 1 dose of study drug, the subject will be included in a summary of adverse events according to the treatment received; otherwise, if the subject is not dosed, then they will be excluded from the summary.
- If safety laboratory results for a participant are missing for any reason at a time point, the subject will be excluded from the calculation of the summary statistics for that time point.

Values for missing safety laboratory data will not be imputed; however, a missing baseline (day 0) result will be replaced with a screening result, if available.

#### **Outliers**

Outliers will be identified during data management and data analysis process, but no sensitivity analyses will be conducted. All data will be included in the data analysis.

#### **Data Handling Conventions and Transformations**

HCV RNA values below the LLOQ for the assay will be set to the lower limit minus 1 for the calculation of summary statistics for the actual HCV RNA values and the change from baseline values by study visit.

For selected analyses, HCV RNA data (IU/mL) will be transformed to the logarithmic (base 10) scale ( $log_{10}$  IU/mL).

#### **Visit Windows**

### **Definition of Study Day**

Study day will be calculated from the date of first dose of study drug administration and derived as follows:

- For post-dose study days: Assessment Date minus First Dose Date + 1
- For days prior to the first dose: Assessment Date minus First Dose Date

The last dose date for an individual study drug will be the end date entered in the Treatment Termination or Drug Administration eCRF.

The last dose date of treatment for a given participant will be defined as the maximum of the last dose dates of individual study drugs in a treatment group, if applicable.

If there are participants for whom the date of last study drug is unknown (lost to follow-up and not able to be contacted), the date of last dose will be estimated using the maximum of non-missing study drug start or stop dates, visit dates, and laboratory collection dates (post-treatment visits and unscheduled visits are not included).

#### **Analysis Windows**

Participant visits might not occur on protocol-specified days. Therefore, for the purposes of analysis, observations will be assigned to analysis windows (**Table 1** and **Table 2**).

In general, the baseline value will be the last non-missing value on or prior to the first dose date of study drug. HCV RNA and safety laboratory data collected up to the last dose date  $+ \le 3$  days are considered to be on-treatment data. HCV RNA and safety laboratory data collected after the last dose date + > 3 days are considered post-treatment data. HCV RNA and safety laboratory data collected after the last dose date + > 3 days will be assigned to the post-treatment follow-up (FU) visits. Visit windows will be calculated from the last dose date (ie, FU Day = collection date minus the last dose date) as shown.

Table 1. On-treatment visit analysis windows

| Nominal visit | | | |
|---------------|-------------|-------------|--------------------|
| NOMINAL VISIT | Nominal day | Lower Limit | <b>Upper Limit</b> |
| Baseline | 1 | NA | 1 |
| Week 2 | 14 | 8 | 21 |
| Week 4 | 28 | 22 | 35 |
| Week 6* | 42 | 36 | 49 |
| Week 8 | 56 | 50 | 63 |
| Week 10 | 70 | 64 | 77 |
| Week 12 | 84 | 78 | <u>&gt;</u> 85 |

<sup>\*</sup>Shortened arm ETR

Table 2. Post-treatment visit analysis windows

| Naminal Ell | HCV RNA | | | Safety Laboratory Data | | |
|---|---|---|---|---|---|---|
| Nominal FU visit | Nominal<br>day | Lower<br>Limit | Upper<br>Limit | Nominal day | Lower<br>Limit | Upper<br>Limit |
| PT week 4 | 28 | 21 | 69 | 28 | 4 | 30 |
| PT week 12 | 84 | 70 | 146 | NA | NA | NA |
| PT week 24 | 168 | 147 | NA | NA | NA | NA |

#### **PARTICIPANT DISPOSITION**

#### Recruitment

The following dates will be presented to define the period of recruitment and follow-up:

- I. first and last participant screened
- II. first and last participant baselined
- III. first and last participant to complete PT week 12

#### **Participant Enrolment and Disposition**

A summary of participant enrolment will be provided- overall and by treatment group (if appropriate). The total number of participants who were screened, enrolled and treated will be depicted by a flowchart (**Figure 2**).

A summary of participant disposition will be provided overall (Table 3).

Reasons for participant exclusion, including screen failure and loss to follow up, will be summarised (**Table 4, Table 5**).

#### **Protocol violations**

Number, proportion, type and reason for any protocol violations will be described (Table 6).

Figure 2. Participant disposition



Table 3. Recruitment and follow-up

| Participant disposition | Total<br>N (%) | Standard<br>arm<br>N(%) | Shortened arm N(%) |
|---|---|---|---|
| Total participants screened, n | | | |
| Participants screened and excluded, n | | | |
| Participants allocated to treatment, N Commenced allocated treatment, n/N (%) Did not commence allocated treatment, n/N (%) | | | |
| Treated Participants | | | |
| Completed allocated treatment course, n (%) Discontinued treatment, n (%) Lost to study follow-up, n (%) | | | |
| Study follow up | | | |
| Completed study follow up, n (%) | | | |
| Did not complete study follow up, n (%) | | | |
| Population for analysis | | | |
| ITT, n | | | |
| mITT, n | | | |
| PP, n | | | |

# Table 4. Reasons for screen failure

| Participant disposition | N (%) |
|-----------------------------------------------------------------|-------|
| Total participants screened, n | |
| Participants screened and excluded, n | |
| Screen fail participants who did not meet eligibility criteria | |
| List reasons (inclusion and exclusion criteria) | |
| Participants who met eligibility criteria but were not enrolled | |
| List reasons for not being enrolled | |
| Lost to follow up | |
| Withdrew consent | |

# Table 5. Reasons for loss to study follow-up

| Study Number | Date of treatment commencement | Date last<br>follow-up | Reason lost to follow-up |
|---|---|---|---|
| Standard Arm | | | |
| Simplified Arm | | | |

# **Table 6. Protocol violations or deviations**

| Protocol violations or deviations | N (%) |
|----------------------------------------------------|-------|
| Total number with protocol violations | |
| Total number with protocol deviations | |
| Violation of study inclusion or exclusion criteria | |
| Enrolment errors | |

#### **BASELINE DATA**

#### **Demographic Data and Baseline Characteristics (Table 7 - 11)**

Demographic and baseline measurements will be summarized using standard descriptive methods. Baseline data will be summarised for the total FAS population and by HCV genotype and HIV serostatus as: number (n) and proportion for categorical parameters; or n, mean and standard deviation (SD), median, Q1, Q3, minimum and maximum for continuous parameters.

Age will be calculated in years at the date of initial study drug administration (baseline).

P values will not be reported for differences between the two groups at baseline, since appropriate randomisation methods will have accounted for this. Any differences identified would be due to chance such that a significant p value would in reality be representative of a type 1 error. Large differences at baseline (more than half a SD for continuous variables or 10% for categorical variables) will be investigated in a sensitivity analysis.

For pre-specified variables and variables only recorded at screening and not at baseline, screening values will be presented in the baseline table.

 Table 7. Participant demographic and clinical enrolment characteristics

| | Total study | Standard | Shortened |
|---|---|---|---|
| <b>Enrolment characteristics</b> | population | Arm | Arm |
| | (n=XXX) | (n=XXX) | (n=xxx) |
| Age, mean (SD) or median (IQR) | | | |
| Gender, n (%) | | | |
| Male | | | |
| Female | | | |
| Transgender | | | |
| Ethnicity, n (%) | | | |
| Caucasian/white | | | |
| Asian | | | |
| Black | | | |
| Other | | | |
| BMI, mean (SD) or median (IQR or range) | | | |
| HCV genotype/subtype, n (%) | | | |
| Genotype 1 | | | |
| 1a | | | |
| 1b | | | |
| 1, not specified | | | |
| Genotype 2 | | | |
| 2a | | | |
| 2b | | | |
| Genotype 3 | | | |
| 3a | | | |
| Genotype 4 | | | |
| Genotype 5 | | | |
| Genotype 6 | | | |
| Genotype mixed | | | |
| Specify | | | |
| Genotype indeterminate | | | |
| HCV RNA, IU/mL | | | |
| Quantitative, mean (SD) or median (IQR or | | | |
| range) | | | |
| Log10, mean (SD) or median (IQR or range) | | | |
| Classification of recent HCV Infection | | | |
| Primary | | | |
| Reinfection | | | |
| Duration of infection, mean (SD) or median | | | |
| (IQR or range) | | | |
| Acute | | | |
| Chronic | | | |

Table 8. Other baseline demographic and socio-economic characteristics

| Variable | Total | Standard arm | Shortened<br>arm |
|---|---|---|---|
| Sexuality, n (%) | | | |
| Source of income, n (%) | | | |
| Highest level of education, n (%) | | | |
| Accommodation, n (%) | | | |
| Rented house/flat; privately owned house/flat; boarding | | | |
| house; hostel; psychiatric home; alcohol/drug treatment | | | |
| residence; shelter/refuge; prison/detention centre; caravan; | | | |
| no usual residence, squat; other | | | |
| Social functioning score, mean (SD) or median (IQR) | | | |
| Who do you live with? | | | |
| Alone; spouse partner; Alone with children; spouse/partner | | | |
| and children; other relatives; friends; | | | |
| friends/parents/relative and children; other | | | |
| Been in prison/juvenile justice, n(%) | | | |
| Ever; last 6 months | | | |
| Clinician determined mode of HCV exposure, n (%) | | | |
| Self-reported mode of HCV exposure, n (%) | | | |
| Injecting drug use/ Transfusion of blood products/ | | | |
| Occupational (needle stick or other exposure)/ Sexual | | | |
| exposure to a known HCV positive person of the same sex/ | | | |
| Sexual exposure to a known HCV positive person of the | | | |
| opposite sex/ Sexual exposure to persons of unknown HCV | | | |
| status of the same sex/ Sexual exposure to persons of | | | |
| unknown HCV status of the opposite sex/ Body piercing/ | | | |
| Tattoos/ Use of recreational drugs (snorting/inhaling)/ | | | |
| Other (please specify) | | | |
| PrEP use in past 6 months (among HIV negative), n(%) | | | |
| Never/ Yes every day/ Yes every week (4-6 days per | | | |
| week)/ Yes every week (1-3 days per week)/ Yes, | | | |
| occasionally (the day or two before or after sex) | | | |
| Screened for STDs in last 12 months, n (%) | | | |
| STD diagnosed in last 12 months prior to HCV diagnosis, | | | |
| n(%) | | | |
| Listing of STDs among those diagnosed | | | |

**Table 9. Participant viral enrolment characteristics** 

| Baseline characteristics | Total study population N=XXX | Standard<br>Arm<br>N=XXX | Shortened<br>Arm<br>N=XXX |
|---|---|---|---|
| HCV | | | |
| ALT (U/L), median (IQR) | | | |
| Peak ALT prior to enrolment | | | |
| ALT at baseline | | | |
| Prior HCV treatment, n (%) | | | |
| Yes | | | |
| (Specify) | | | |
| Response to prior HCV treatment, n/total "Yes" (%) | | | |
| Non-response | | | |
| Breakthrough | | | |
| Relapse | | | |
| Other (specify) | | | |
| Fibroscan performed, n (%) | | | |
| Valid Fibroscan, n/N (%) | | | |
| Median liver stiffness measurement (Fibroscan®), kPa | | | |
| (IQR) | | | |
| (in those with <b>valid</b> Fibroscan result only) | | | |
| HIV | | | |
| HIV infection, n (%) | | | |
| CD4 count (10 <sup>6</sup> /L), median (IQR) | | | |
| HIV VL ≤50 at screening, n (%) | | | |
| On cART, n (%) | | | |
| HBV | | | |
| HBsAg positive, n (%) | | | |
| HBcAb positive, n (%) | | | |
| HsAb >10 IU/ml, n (%) | | | |
| HBV DNA detected, n (%) | | | |
| NA therapy for HBV, n (%) | | | |

Abbreviations: Combination antiretroviral therapy (cART); nucleos(t)ide analogue (NA)

Table 10. History of substance use at enrolment

| Substance use characteristics | Total<br>N= | Standard<br>Arm<br>N= | Shortened Arm<br>N= |
|---|---|---|---|
| Injecting drug use, n (%) | | | |
| Ever | | | |
| Recent <sup>a</sup> | | | |
| Current <sup>a</sup> | | | |
| In those reporting injecting drug use: | | | |
| Age at first injecting, median (range) | | | |
| Last injected within 30 days, n (%) | | | |
| Last injected between 1-6 months ago, n (%) | | | |
| Last injected >6 months ago, n (%) | | | |
| If injected in the previous 1 month, frequency (n, %): | | | |
| >3x most days | | | |
| .2-3x most days | | | |
| Daily | | | |
| More than weekly, but less than daily | | | |
| Less than weekly | | | |
| Drug injected most in last month, n (%) <sup>b</sup> | | | |
| Heroine | | | |
| Cocaine | | | |
| Methamphetamines | | | |
| Other opiates | | | |
| Benzodiazepines | | | |
| Opioid substitution therapy, n (%) | | | |
| Never | | | |
| Ever | | | |
| Cot currently | | | |
| Current | | | |
| Alcohol use, n (%) <sup>c</sup> | | | |
| None | | | |
| Frequency n (%) | | | |
| Monthly or less; | | | |
| 2 - 4 times/month | | | |
| 2 -3 times/week | | | |
| 4 or more times/week | | | |
| Standard drinks per day n (%) | | | |
| Mean (SD); Median (IQR) | | | |
| Frequency of Six or more standard drinks on one occasion n (%) | | | |
| Never, less than monthly, monthly, weekly, almost daily/ daily | | | |
| AUDIT C Score n (%) | | | |
| Number identified as hazardous drinkers n (%) | | | |

<sup>a</sup> Recent injecting drug use refers to use within 6 month of screening, and Current injecting within the past month; <sup>b</sup> other drugs not listed that will also be summarised: Oxycodone, methadone, buprenorphine, fentanyl, steroids, LSD or other hallucinogens, Ecstasy; <sup>c</sup> One standard drink = 10 grams of alcohol

Table 11. Of syringe sharing among Injecting drug users

| | Total | Standard | Shortened Arn |
|---|---|---|---|
| Syringe sharing use characteristics <sup>a</sup> | N= | Arm | N= |
| | | N= | |
| Use of NEW sterile needle and syringe in last month, n (%) | | | |
| All injections | | | |
| Most of the time <sup>a</sup> | | | |
| Half of the time | | | |
| Some of the time | | | |
| Not in the last month | | | |
| How many times in last month used a needled/syringe after someone | | | |
| else, n (%) | | | |
| None | | | |
| One time | | | |
| Two times | | | |
| 3 – 5 times | | | |
| More than 5 times | | | |
| Who did you share with?, n (%) | | | |
| No-one | | | |
| Regular sex partner | | | |
| Casual sex partner | | | |
| Close friends | | | |
| Acquaintance | | | |
| Other | | | |
| How many times in last month has someone used a needled/syringe | | | |
| after you, n (%) | | | |
| None | | | |
| One time | | | |
| Two times | | | |
| 3 – 5 times | | | |
| More than 5 times | | | |
| Who were these people that shared after you?, n (%) | | | |
| No-one | | | |
| Regular sex partner | | | |

Casual sex partner Close friends Acquaintance

Other

<sup>&</sup>lt;sup>a</sup> Denominator – those reporting injecting drug use in last month

# **STUDY ENDPOINTS**

Table 12. Study endpoints and outcomes

| | | I |
|---|---|---|
| Primary endpoint | Non-inferiority of simplified on- | Included in primary analysis |
| | treatment monitoring to standard on- | |
| | treatment monitoring (ITT population) | |
| Secondary endpoints | Non-inferiority of simplified on- | Included in primary analysis |
| | treatment monitoring to standard on- | |
| | treatment monitoring (mITT population) | |
| | Non-inferiority of simplified on- | Included in primary analysis |
| | treatment monitoring to standard on- | |
| | treatment monitoring (PP population) | |
| | Treatment response: ETR, SVR4, SVR24; | Included in primary analysis |
| | HCV RNA below the level of | |
| | quantification through 2 years post | |
| | treatment | |
| | Adverse events | Included in primary analysis |
| | On-treatment adherence | Included in primary analysis |
| | Early treatment discontinuation | Included in primary analysis |
| | Relapse and reinfection | Included in primary analysis |
| | Resistance associated substitutions (RAS) | Included in primary analysis |
| | for people who have failed treatment | , , , |
| | Laboratory abnormalities | Included in primary analysis |
| | Change in HIV RNA and CD4 (on | Included in primary analysis |
| | treatment and end of treatment) | , , , |
| | , | |
| | | Included in primary analysis |
| Additional pre- | Factors associated with on treatment | Included in primary analysis |
| specified outcomes | efficacy (only if SVR12 is low) | moraded in primary disarysis |
| | Factors associated with sub-optimal | |
| | adherence | |
| | Factors associated with re-infection | Not included in primary analysis |
| | Tactors associated with re-in-consti | The mercada in primary anarysis |
| | To evaluate the impact of treatment on | Not included in primary analysis |
| | illicit drug use, injecting behaviour and | Troc meradea in primary analysis |
| | sexual risk-taking behaviour (behavioural | |
| | survey) during treatment | |
| | To evaluate patient interest and attitudes | Not included in primary analysis |
| | towards long acting parenteral hepatitis C | |
| | therapy (Long-Acting Hepatitis C Therapy | |
| | Questionnaire) | |
| | | L |

#### **Primary efficacy endpoint**

The proportion of participants with HCV RNA below the level of quantitation (target not detected [TND] or target detected, not quantifiable [TDnq]) at 12 weeks post end of treatment (SVR12)

The primary analysis will compare randomised treatment groups on an ITT basis including all available data. The primary endpoint, SVR12, will be calculated for each patient based on all available data. Treatment arms will be regarded as non-inferior if the difference in proportion between regimens has a lower limit greater than -12%. Secondary analyses will compare randomised treatment groups based on available data (per protocol).

#### Secondary efficacy endpoints

- Virological endpoints
  - The proportion of treated participants with:
    - ETR (defined as undetectable plasma HCV RNA at the end of treatment)
    - SVR4 (defined as undetectable plasma HCV RNA at post-treatment week 4)

For virological endpoints, the point estimates and 95% exact confidence intervals will be reported by study arm, by HCV genotype and by HIV serostatus.

#### Virological endpoints (Table 13 and 14)

The presence of HCV RNA will be assessed at all scheduled clinic study visits using Aptima HCV Quant Dx assay, version 2.15.5 (lower limit of quantitation [LLoQ] 10IU/mL; Hologic, Inc., Marlborough, MA, USA), with centralised testing performed at St Vincent's Centre for Applied Medical Research (Sydney, NSW, Australia).

Proportions and 95% confidence intervals will be reported for both the primary and secondary virological endpoints. Virological endpoints will be assessed in the ITT, mITT and PP populations, with results stratified by HCV genotype/subtype and HIV serostatus.

Factors associated with treatment outcome in the ITT population will be evaluated by univariate analysis. Variables assessed will include but are not limited to: demographic factors (age, gender); virological factors (baseline HCV RNA, genotype 1 subtype, duration of HCV infection); risk behaviors (injecting drug use, sexual behavior, mode of HCV acquisition); HIV co-infection; treatment factors (adherence).

#### **Primary safety endpoints**

The primary safety endpoints are:

- Proportion of participants with common adverse events (reported by greater than 5% of the study population);
- Proportion of participants with at least one severe or potentially life threatening (grade 3 or 4) adverse event;

#### Adherence

80% adherence: Defined as the receipt of >80% of scheduled doses. 90% adherence: Defined as the receipt of >90% of scheduled doses. 100% adherence: Defined as the receipt of 100% of scheduled doses.

On-treatment adherence will be calculated by subtracting the number of missed doses from the total number of doses of scheduled treatment and dividing by the total intended therapy duration. This measures the proportion of doses received from the time that treatment was initiated until treatment was discontinued or completed.

Table 13. Primary and secondary efficacy endpoints – (ITT)

| Efficacy | Arm A Standard treatment (N=XX) | Arm B<br>Shortened<br>treatment<br>(N=XX) | Difference<br>between arms<br>(95% CI) | P value |
|---|---|---|---|---|
| ETR, n (%) | | | | |
| SVR 4, n (%) | | | | |
| SVR 12, n (%) | | | | |
| Non-response | | | | |
| Relapse | | | | |
| Reinfection | | | | |
| Lost to follow up | | | | |
| SVR 24, n (%) | | | | |
| Virologic failure, n (%) On-treatment failure (non-response, breakthrough) Relapse* | | | NA | |

<sup>\*</sup>relapse definition:

Analysis tables will also be presented for the mITT, and PP populations

Table 14. SVR12 in participant subgroups, ITT population

| Subgroup | Standard tx arm<br>n/N (%; 95% CI) | Shortened tx arm<br>n/N (%; 95% CI) |
|---|---|---|
| HCV mono-infection | | |
| HIV/HCV co-infection | | |
| Genotype 1 | | |
| Genotype 1a | | |
| Genotype 1b | | |
| Genotype 2 | | |
| Genotype 3 | | |
| Genotype 4 | | |
| Genotype 5 | | |
| Genotype 6 | | |

# Other secondary outpoints

Table 15: Primary reason for premature discontinuation of study drug

| Reason for premature discontinuation, n (%) | Standard tx arm<br>(n=XXX) | Shortened tx arm (n=XXX) |
|---|---|---|
| Adverse event | | |
| Non-compliance | | |
| Withdrawal of consent | | |
| Loss to follow up | | |
| Other | | |
| Specify - list | | |

# Table 16: Reinfection by SVR12

| | N | % | 95% CI |
|---------------|---|---|--------|
| Standard Arm | | | |
| Shortened Arm | | | |

# Table 17: Relapse by SVR12

| | N | % | 95% CI |
|---------------|---|---|--------|
| Standard Arm | | | |
| Shortened Arm | | | |

Table 18. Prevalence of polymorphisms in NS5B and NS5A at baseline

| Polymorphism, n (%) | Total study population N=XXX | Standard duration<br>arm<br>N=XXX | Shortened<br>duration arm<br>N=XXX |
|---|---|---|---|
| Any NS5B | N | N | N |
| [Specify] | | | |
| Any NS5A | N | N | N |
| M28G/S/T | | | |
| L31F/I/M/P/V | | | |
| P32A/L/Q/R | | | |
| A/C92K/T | | | |
| Y93D/H/N/R/S/W | | | |

Baseline polymorphisms detected by Sanger sequencing at the following amino acid positions:

NS5A: 28, 31, 32, 92, 93

Table 19. NS5B and NS5A polymorphisms at baseline and virologic failure

| Subject ID | Genotype and | Virologic failure | NS5B V | ariants | NS5A v | ariants |
|---|---|---|---|---|---|---|
| Subject 1D | subtype | virologic failure | Baseline | Failure | Baseline | Failure |
| Standard treatme | Standard treatment duration (12 weeks), n=XXX | | | | | |
| Shortened treatm | Shortened treatment duration (6 weeks), n=XXX | | | | | |

Table 19. Characteristics of participants with virological failure

| | Genotype and | | Genetic distance % <sup>1</sup> | | Baseline<br>HCV | |
|---|---|---|---|---|---|---|
| Subject ID | subtype | Virologic failure | Core-E2 <sup>1</sup> | NS5A | RNA<br>(log <sub>10</sub> ) | Adherent <sup>2</sup> |
| Standard treatment duration (12 weeks), n=XXX | | | | | | |
| Shortened treatment duration (6 weeks), n=XXX | | | | | | |

<sup>1.</sup> Reported genetic distance % for Core-E2 and NS5A was the comparison between sequences at baseline and post-treatment week 12. Cut-off for homologous virus was <4% for Core-E2 and X% for NS5A.

Table 21. On treatment adherence

| | N | % | 95% CI |
|----------------|---|---|--------|
| 80% adherence | | | |
| Standard Arm | | | |
| Shortened Arm | | | |
| 90% adherence | | | |
| Standard Arm | | | |
| Shortened Arm | | | |
| 100% adherence | | | |
| Standard Arm | | | |
| Shortened Arm | | | |

<sup>2.</sup> Adherence was defined as receipt of ≥95% of the prescribed treatment course

#### **SAFETY ANALYSES**

All participants who receive at least one dose of study drug will be included in the safety analyses. Safety analyses will be performed overall and by treatment arm. Safety will be evaluated by assessment of clinical laboratory tests at various time points during the study, and by the documentation of AEs.

All safety data collected on or after the first dose of study drug administration up to 30 days after the last dose of study drug will be summarised.

#### **Extent of Exposure**

A participant's extent of exposure to study drug will be generated from the study drug administration page of the eCRF.

#### **Adverse Events**

Clinical and laboratory AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, insert version). System organ class (SOC), high level group term (HLGT), high level term (HLT), preferred term (PT), and lower level term (LLT) will be provided.

Events will be summarised on the basis of the date of onset for the event.

A treatment-emergent AE (TEAE) will be defined as:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
- Any AEs leading to premature discontinuation of study drug

#### **Adverse Event Severity**

Adverse events are graded by the investigator as mild (Grade 1), moderate (Grade 2), severe (Grade 3), or life-threatening (Grade 4) according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings, and the most severe will be considered (for sorting purpose only) in data presented. For example, if an adverse event of the same type (PT) is listed more than once for an individual, the highest grade will be used to summarise severity.

# Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" ("Possibly related" or "Probably related") on the AE CRF to the question of "Related to Study Treatment." Events for which the investigator did not record the relationship to study drug will be considered to be related to study drug for summary purposes.

#### **Summaries of Adverse Events and Deaths**

The number and percentage of participants overall and in each arm with treatment-emergent adverse events will be tabulated by primary MedDRA System Organ Class (SOC) and preferred term (PT). The tabulation of the number of participants with treatment-emergent adverse events by severity grade and relationship to study drug also will be provided.

Participants reporting more than one adverse event for a given MedDRA PT will be counted only once for that term using the most severe grade for the severity grade table and the most related for

the relationship to study drug tables. Participants reporting more than one type of event within a SOC will be counted only once for that SOC, but both PTs will be listed.

Summaries of treatment-emergent AEs (by SOC and PT) will be provided for the following:

- All TEAEs
- TEAEs of Grade 3 or above
- All treatment-related TEAEs
- Treatment-related TEAEs of Grade 3 or above
- All SAEs (including death)
- All treatment-related SAEs
- All TEAEs leading to premature discontinuation of the study drug
- TEAEs that occurred in at least 5% of subjects within any treatment group

Adverse event summaries will provide the number and percentage of subjects with treatmentemergent AEs by SOC and PT, divided by treatment group.

Adverse events will be summarised and listed first in alphabetic order of SOC and then by PT in order of descending incidence of the pooled treatment groups within each SOC.

In summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in a participant during the study.

#### Serious adverse events (SAE)

The proportion of participants with at least one SAE will be reported overall. Serious adverse events will be summarized and relationship between the SAE and study drug will be detailed

#### **Laboratory Evaluation**

Selected laboratory data will be summarised (n, mean, SD, median, IQR, range) by study visit along with the corresponding change from Baseline/Day 1 to Post Treatment Week 12.

Depending on sample distribution, parametric or non-parametric tests can be used to compare the change in biochemical and haematological indicators over time.

The NIH DAIDS AE Grading Table Version 2.0- November 2014 will be used to grade severity.

Table 22. Safety parameters – adverse events and treatment discontinuation

| Adverse events | Safety analysis set<br>(N=XX) |
|---|---|
| Participants reporting any AE up to 30 days after last dose, n (%) | |
| Grades 1-2, n (%) | |
| Grade 3, n (%) | |
| Grade 4, n (%) | |
| Participants reporting treatment-related AE up to 30 days after | |
| last dose, n (%) | |
| Grades 1-2, n (%) | |
| Grade 3, n (%) | |
| Grade 4, n (%) | |
| Serious adverse event, n (%) | |
| Treatment-related serious adverse event, n (%) | |
| Treatment discontinuation due to adverse event, n (%) | |
| Death, n (%) | |
| Adverse events | |
| Common (>10% of study population), n (%) | |
| Specify (list) | |

# Table 23. Listing of serious adverse events

| Study<br>Arm | Date<br>Onset | Date<br>resolved | Diagnosis or event description | SAE<br>criteria‡ | <b>Outcome</b> § | Relationship to study drug |
|---|---|---|---|---|---|---|
| Standard | | | | | | |
| Shortened | | | | | | |

<sup>‡</sup> Death, hospitalised, life threatening, medically important, congenital anomaly, disability

Table 24. Serious adverse events summary

| SAE – event summary | All<br>N=XXX | Treatment<br>arm 1<br>N=XXX | Treatment<br>arm 2<br>N=XXX |
|---|---|---|---|
| N of participants experiencing any treatment-emergent SAE by | | | |
| MedDRA SOC and Preferred Term, n (%) | | | |
| SOC (alphabetical order) | | | |
| List PT | | | |

<sup>§</sup> Recovered, Improved, Unchanged, Worsened, Unknown, Died

# **Laboratory Evaluation**

Selected laboratory data will be summarised (n, mean, SD, median, IQR, range) by study visit along with the corresponding change from Baseline/Day 1.

**Table 25. Summary table for key laboratory evaluations** 

| Lab parameter | N | Mean | SD | Min | Q1 | Median | Q3 | Max |
|---------------|---|------|----|-----|----|--------|----|-----|
| ALT | | | | | | | | |
| AST | | | | | | | | |
| Glucose | | | | | | | | |
| ALP | | | | | | | | |
| Albumin | | | | | | | | |
| Creatinine | | | | | | | | |
| Haemoglobin | | | | | | | | |
| WBC | | | | | | | | |
| Neutrophils | | | | | | | | |
| Platelets | | | | | | | | |
| Bilirubin | | | | | | | | |

<sup>\*</sup>table will be further stratified by Arm and study weeks (Screening, baseline, Week 4, ETR, SVR4)

Table 26. HIV patients only – changes in HIV viral load and CD4 cell count

| Parameter | Standard Arm | Shortened arm |
|-----------------------------|--------------|---------------|
| HIV viral load (<20 copies) | N (%) | N (%) |
| Screening | | |
| Baseline | | |
| Week 4 | | |
| SVR12 | | |
| Change in CD4 cell count | Mean (SD) | Mean (SD) |
| Screening | | |
| Baseline | | |
| SVR12 | | |

Table 27. Listing of HIV patients with VL > 200 copies at any timepoint, by treatment arm

| Study Arm | Study ID | Week first VL >200 copies/mL |
|-----------|----------|------------------------------|
| Standard | | |
| Shortened | | |

Table 28. Grading of severity of laboratory measures

| Laboratory evaluation | Standard Arm<br>(N=XX) | Shortened Arm<br>(N=XX) |
|---|---|---|
| Haematological parameters | | |
| Baseline Hb, g/L (mean, SD) | | |
| Change in Hb at post-treatment week 12, g/L (mean, SD) | | |
| Haemoglobin <sup>#</sup> , n (%) | | |
| Grade 2 | | |
| Grade 3 | | |
| Grade 4 | | |
| Biochemical parameters | | 1 |
| Baseline ALT, U/L (mean, SD) | | |
| ALT, n (%) | | |
| Grade 2 (3-5x ULN) | | |
| Grade ≥3 (>5x ULN) | | |
| Change in ALT at post-treatment week 12, g/L (mean, SD) | | |
| Baseline AST, U/L (mean, SD) | | |
| AST, n (%) | | |
| Grade 2 (3-5x ULN) | | |
| Grade ≥3 (>5x ULN) | | |
| Change in AST at post-treatment week 12, g/L (mean, SD) | | |
| Baseline total bilirubin, mg/dl or mmol/L (mean, SD) | | |
| Total bilirubin *, n (%) | | |
| >2.5-3.0 mg/dl (43 – 51 mmol/L) | | |
| >3.0 mg/dl (>51 mmol/L) | | |
| Change in bilirubin at post-treatment week 12, g/L | | |
| (mean, SD) | | |

<sup>&</sup>lt;sup>#</sup> At any time during treatment and up to 30 days post; each participant should only be included once

<sup>-</sup> record most severe grade of anaemia for each participant

<sup>\*</sup>At any time during treatment and up to 30 days post; add footnote, if bilirubin elevated at screening/baseline